CLINICAL TRIAL: NCT05792722
Title: A Prospective, Randomized Trial Comparing Prostate Capsule-sparing and Nerve-sparing Radical Cystectomy in Patients With Bladder Cancer
Brief Title: Evaluating Safety and Efficacy of Prostate-sparing Radical Cystectomy
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRB00345549
Record Dates: First submitted 2023-03-16; First posted 2023-03-31 (Actual); Last update posted 2025-11-18 (Actual); Status verified 2025-11

CONDITIONS: Bladder Cancer
Keywords: Radical Cystectomy; Prostate Capsule-Sparing Cystectomy; Nerve-Sparing Cystectomy; Male
MeSH Terms: conditions — Urinary Bladder Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Prostate Capsule-Sparing Radical Cystectomy (Other): Patients randomized to this arm will receive the prostate capsule-sparing surgery performed in the form of standard simple prostatectomy. Patients will also have a cystectomy with one of the following urinary diversions: ileal conduit, Indiana Pouch, or orthotopic neobladder.
  Interventions: Procedure: Prostate capsule-sparing radical cystectomy
- Nerve-Sparing Radical Cystectomy (Other): Patients randomized to this arm will receive the nerve-sparing surgery will be performed in the form of the standard nerve-sparing radical prostatectomy. Patients will also have a cystectomy with one of the following urinary diversions: ileal conduit, Indiana Pouch, or orthotopic neobladder.
  Interventions: Procedure: Nerve sparing radical cystectomy

INTERVENTIONS:
Procedure: Prostate capsule-sparing radical cystectomy — Patients randomized to this arm will receive the prostate capsule-sparing surgery performed in the form of standard simple prostatectomy. Patients will also have a cystectomy with one of the following urinary diversions: ileal conduit, Indiana Pouch, or orthotopic neobladder.
  Arms: Prostate Capsule-Sparing Radical Cystectomy
Procedure: Nerve sparing radical cystectomy — Patients randomized to this arm will receive the nerve-sparing surgery will be performed in the form of the standard nerve-sparing radical prostatectomy. Patients will also have a cystectomy with one of the following urinary diversions: ileal conduit, Indiana Pouch, or orthotopic neobladder.
  Arms: Nerve-Sparing Radical Cystectomy

SUMMARY:
The purpose of this clinical trial is to determine if prostate-capsule-sparing cystectomy improves functional outcomes without comprising oncologic outcomes in male patients receiving a radical cystectomy. Patients will be randomized to one of two groups: prostate capsule-sparing radical cystectomy or nerve-sparing radical cystectomy. Patients will be monitored following standard of care guidelines and clinical data will be collected. Patients in both groups will be asked to complete an erectile function questionnaire at multiple timepoints. Patients who receive an orthotopic neobladder will be asked to complete a questionnaire to monitor urinary function at multiple timepoints. Patient adverse events will be monitored to ensure patients safety.

DETAILED DESCRIPTION:
The purpose of this study is to determine if prostate capsule-sparing cystectomy improves functional outcomes without compromising the oncologic outcomes in patients with bladder cancer. The comparison arm will be patients undergoing nerve-sparing radical cystectomy. Participants will be randomized to receive either a nerve-sparing radical cystectomy or a prostate capsule-sparing radical cystectomy. Patients will be monitored following standard of care guidelines every 3-months post-operatively up to and including 24 months post-operatively. As part of standard of care post-operative follow-up patients will have routine history and physical exams, urine cytology, urine culture, Complete Blood Count (CBC), Comprehensive Metabolic Panel (CMP), and Prostate Specific Antigen (PSA). Standard of Care diagnostic imaging will also occur. The Sexual Health Inventory for Men (SHIM) Questionnaire will be given to patients 6-weeks post-operatively and every 3-months post-operatively up to and including 24-months post-operatively. To measure urinary function in patients who receive orthotopic neobladder, the Validated Pad Questionnaire will be given 6-weeks post-operatively and every 3-months post-operatively up to and including 24-months post operatively. Adverse Events will be monitored in both groups as defined by the CTCAE 5.0 guidelines.

ELIGIBILITY:
Inclusion Criteria:

* Subjects with pathologically confirmed bladder cancer scheduled for radical cystectomy
* Variant histologies of bladder cancer permitted
* Neoadjuvant therapy permitted
* Age > 18 years old
* Ability to understand and willingness to sign a written informed consent document

Exclusion Criteria:

* Patients that are not candidates for cystectomy
* Moderate to severe erectile dysfunction with SHIM score <17
* Bladder cancer with bladder neck or prostatic involvement, including cancer in the prostatic urethra
* Prior pelvic radiation
* Confirmed prostate cancer:
* Patients with abnormal Digital rectal exam (DRE), PSA >3 or Prostate Imaging Reporting & Data System (PIRADS) 4 lesions on prostate Multiparametric MRI (mpMRI) will undergo prostate biopsy to rule out prostate cancer
* Increased genetic risk of prostate cancer per National Comprehensive Cancer Network (NCCN) guidelines:
* ≥1 first-, second-, or third-degree relative with: breast cancer at age ≤50 y, colorectal or endometrial cancer at age ≤50 y, male breast cancer at any age, ovarian cancer at any age, exocrine pancreatic cancer at any age, metastatic, regional, very-high-risk, high-risk prostate cancer at any age
* ≥1 first-degree relative (father or brother) with: prostate cancer at age ≤60 y
* ≥2 first-, second-, or third-degree relatives with: breast cancer at any age, prostate cancer at any age
* ≥3 first- or second-degree relatives with: Lynch syndrome-related cancers, especially if diagnosed
* Patients with Lynch syndrome

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2023-10-25 (Actual); Primary Completion 2028-07 (Estimated); Study Completion 2029-07 (Estimated)

PRIMARY OUTCOMES:
Change in Functional Outcomes as assessed by the Sexual Health Inventory for Men (SHIM) | Baseline, 6 weeks-post operatively, 3-months post-operatively, 6-months post-operatively, 9-months post-operatively, 12-months post-operatively, 15-months post-operatively, 18-months post-operatively, 21-months post-operatively, 24-months post-op
  Comparison of functional outcomes focusing on preservation of erectile function in patients undergoing cystectomy for bladder cancer. Functional Outcomes will be measured by the Sexual Health Inventory for Men (SHIM) Questionnaire. The Sexual Health Inventory for Men defines the following ranges of Erectile Dysfunction (ED): 1-7 is Severe ED, 8-11 Moderate ED, 12-16 Mild to Moderate ED, and 17 to 21 is Mild ED.

SECONDARY OUTCOMES:
Change in urinary function in patients with orthotopic neobladder as assessed by the Validated Pad Questionnaire | Baseline, 6 weeks-post operatively, 3-months post-operatively, 6-months post-operatively, 9-months post-operatively, 12-months post-operatively, 15-months post-operatively, 18-months post-operatively, 21-months post-operatively , 24-months post-op
  Urinary function in patient with orthotopic neobladder urinary diversions measured using the Validated Pad Questionnaire. The Validated Pad questionnaire will be used to determine the percentage of patients utilizing 1 to 2 pads versus 2 or more pads for night and day, respectively.
Change in overall patient survival | Baseline, 6 weeks-post operatively, 3-months post-operatively, 6-months post-operatively, 9-months post-operatively, 12-months post-operatively, 15-months post-operatively, 18-months post-operatively, 21-months post-operatively, 24-months post-op
  Comparing the overall survival of patients in both arms of the study
Change in disease specific status | Baseline, 6 weeks-post operatively, 3-months post-operatively, 6-months post-operatively, 9-months post-operatively, 12-months post-operatively, 15-months post-operatively, 18-months post-operatively, 21-months post-operatively, 24-months post-op
  Comparing the status of disease specific in both arms of the study
Soft tissue surgical margin rate as assessed by pathology | Up to 4-weeks after surgical intervention
  Pathologists will examine the soft tissue surgical margin rate to determine positive or negative soft tissue surgical margin.
Safety as assessed by adverse events experienced by study participants | Up to 24-months post-operative
  Comparing the differences in adverse events (grades 2-5) as experienced by the participants of in each study arm. The grading of adverse events are defined by the CTCAE 5.0 guidelines.

CONTACTS AND LOCATIONS:
Overall Officials: Armine Smith, MD, Principal Investigator — Johns Hopkins University
Locations (2):
- United States (2):
  - Sibley Memorial Hospital, Washington D.C., District of Columbia
  - Johns Hopkins Hospital, Baltimore, Maryland